CLINICAL TRIAL: NCT07198490
Title: Construction of a Prognostic Model for Severe Brain-Injured Patients Based on Integrated Metabolic-Neurological Monitoring: A Prospective Observational Study
Brief Title: Construction of a Prognostic Model for Severe Brain-Injured Patients Based on Integrated Metabolic-Neurological Monitoring
Acronym: CPM-Brain
Status: Not yet recruiting | Type: Observational
Sponsor: Xingui Dai (Other)
Responsible Party: Sponsor-Investigator, Xingui Dai, The department of Critical Care Medicine, First People's Hospital of Chenzhou
Organization: First People's Hospital of Chenzhou (Other)
Other Study IDs: Chenzhou People's Hospital
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Brain Injuries
Keywords: continuous glucose monitoring,Neurological Multimodal Monitoring,Brain Injury,Intensive Care Unit
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational cohort study aimed at constructing a machine learning-based prognostic model for severe brain-injured patients. The study will synchronously collect continuous glucose monitoring (CGM), electroencephalography (EEG), near-infrared spectroscopy (fNIRS), transcranial Doppler (TCD), and serum neuronal injury biomarkers (NSE, S100β) within 72 hours post-injury. The goal is to investigate the correlation between glycemic variability (GV) and neurological function and to develop an integrated model for early prediction of 3-6 month neurological outcomes (GOSE score).

DETAILED DESCRIPTION:
This study intends to enroll 50 adult patients with brain injury admitted to the ICU. Multimodal monitoring data will be collected prospectively. Machine learning algorithms will be used to integrate the data and build a predictive model. The study will test whether integrated metabolic-neurological monitoring outperforms traditional single-parameter prognostic methods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe TBI, large-volume stroke, or HIE
* Expected ICU stay >72 hours
* Informed consent from legal surrogate

Exclusion Criteria:

* Terminal organ failure
* Pre-existing severe neurological disease
* Skull defect preventing monitoring
* Pregnancy or lactation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (≥18 years old) admitted to the Intensive Care Unit (ICU) of Chenzhou First People's Hospital with a diagnosis of brain injury. This includes patients with:Severe Traumatic Brain Injury (TBI), Expected ICU stay >72 hours,Informed consent from legal surrogate.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extended (GOSE) | 3 and 6 months
  Neurological outcome at 3 and 6 months assessed by Glasgow Outcome Scale Extended (GOSE)

SECONDARY OUTCOMES:
28 days mortality | 28 days
  all cause mortality at days 28

REFERENCES:
- [Background] Jones S, Schwartzbauer G, Jia X. Brain Monitoring in Critically Neurologically Impaired Patients. Int J Mol Sci. 2016 Dec 27;18(1):43. doi: 10.3390/ijms18010043. PMID 28035993
- [Background] Miller C, Armonda R; Participants in the International Multi-disciplinary Consensus Conference on Multimodality Monitoring. Monitoring of cerebral blood flow and ischemia in the critically ill. Neurocrit Care. 2014 Dec;21 Suppl 2:S121-8. doi: 10.1007/s12028-014-0021-9. PMID 25208667
- [Result] Gandee R, Miller C. Multimodality Monitoring: Toward Improved Outcomes. Semin Respir Crit Care Med. 2017 Dec;38(6):785-792. doi: 10.1055/s-0037-1608774. Epub 2017 Dec 20. PMID 29262436